CLINICAL TRIAL: NCT06401616
Title: Anticoagulant Therapy in Patients With Atrial Fibrillation After Surgical Left Atrial Appendage Closure: a Randomized Non-inferiority Trial (The ATLAAC Trial)
Brief Title: Can Patients With Atrial Fibrillation Safely Discontinue Anticoagulant Therapy After Cardiac Surgery? (ATLAAC)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Gødstrup Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Population Health Research Institute (Other); Region of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-502986-92-00; 2022-502986-92-00 (Other: EU-CT)
Record Dates: First submitted 2024-03-05; First posted 2024-05-07 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Absent; Anticoagulant Adverse Reaction
Keywords: Atrial fibrillation; Anticoagulant treatment; Surgical left atrial appendage closure; surgical left atrial appendage occlusion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either continue or discontinue oral anticoagulant therapy
Who Masked: Outcomes Assessor
Masking Description: Blinding of patients and physicians is not possible due to different types of oral anticoagulant therapy within the same interventional arm and the need for continuous monitoring of treatment with warfarin.However, since the primary outcome is not a subjectively reported outcome, lack of blinding presents less risk of bias.
  The investigators responsible for data collection and the Endpoint Adjudication Committee will be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discontinue OAC (Experimental): OAC stopped for the duration of the trial
  Interventions: Drug: OAC will be discontinued for the duration of the trial
- Continue OAC (No Intervention): OAC continued for the duration of the trial

INTERVENTIONS:
Drug: OAC will be discontinued for the duration of the trial — Discontinuation of warfarin, dabigatran, rivaroxaban, apixaban or edoxaban
  Arms: Discontinue OAC

SUMMARY:
Left atrial appendage (LAA) closure has become a frequent addition to oral anticoagulation in patients with atrial fibrillation who undergo cardiac surgery. The procedure significantly reduces the risk of stroke and systemic embolism, which may render anticoagulation unnecessary or even harmful when considering the associated increased risk of bleeding. A clinical trial to address the need for anticoagulation after LAA closure is needed.

The ATLAAC trial will enroll 1220 patients with atrial fibrillation who have previously undergone surgical LAA closure. Patients will undergo a cardiac CT-scan to determine if LAA closure was successful and patients with successful closure will be randomized to continue or discontinue anticoagulation. The trial will assess the risk of ischemic stroke, peripheral arterial embolism, and major bleeding during the randomized intervention

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Previously undergone any type of cardiac surgical procedure including any type of surgical LAA closure (use of any of the following techniques; amputation and suture closure, stapler closure, non-amputating suture closure or closure with an approved surgical occlusion device (e.g. AtriClip)) according to the NationalPatient Register (NPR), the Danish Heart Registry (DHR) or the Western Danish Heart Registry (WDHR) from January 1st 2010 til 3 months prior to inclusion in the project.
* Documented history of paroxysmal, persistent, or permanent atrial fibrillation or atrial flutter according to the electronic patient record
* Informed consent

Exclusion Criteria:

* Not receiving OAC (warfarin/DOAC)
* Patient specific conditions requiring OAC (e.g.mechanical valve, previous pulmonary embolism)
* Renal impairment (estimated glomerular filtration rate < 30)
* Allergy to contrast media
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ischemic strokes, peripheral arterial embolisms and major bleedings | After 128 primary outcome events (approx 4 years)
  Composite endpoint including the occurrence of ischemic stroke, peripheral arterial embolism, and major bleeding (ISTH definition)

SECONDARY OUTCOMES:
Severity of stroke | After 128 primary outcome events (approx 4 years)
  According to Scandinavian Stroke Scale (0-58), lower scores mean worse outcomes
Occurence of transient ischemic attacks | After 128 primary outcome events (approx 4 years)
Occurence of all-cause stroke | After 128 primary outcome events (approx 4 years)
Rate of all-cause mortality | After 128 primary outcome events (approx 4 years)
Rate of cardiovascular mortality | After 128 primary outcome events (approx 4 years)
Occurence of minor bleeding | After 128 primary outcome events (approx 4 years)
  All types of bleeding leading to hospital contact
Number of participants who receive blood transfusion | After 128 primary outcome events (approx 4 years)
Occurence of myocardial infarction | After 128 primary outcome events (approx 4 years)
Occurence of deep venous thrombosis | After 128 primary outcome events (approx 4 years)
Occurence of pulmonary embolism | After 128 primary outcome events (approx 4 years)
Health-related Quality of Life (HRQOL) | Baseline (day 0) and 1 and 2 years after inclusion
  EQ-5D-5L (EuroQol-5 Dimensions-5 Levels) score to evaluate generic HRQOL (0-100). Higher scores mean better quality of life.
Patient-reported satisfaction with overall medical treatment | Baseline (day 0) and 1 and 2 years after inclusion
  Treatment Satisfaction Questionnaire (TSQM) to evaluate satisfaction related to their overall medical treatment. TSQM scoring is by domain and each domain score is computed by summing the individual TSQM items in each domain and then transforming the composite score into a value ranging from 0 to 100. Higher scores indicate higher patient satisfaction with medication.
Patient-reported satisfaction with anticoagulant treatment | Baseline (day 0) after inclusion
  Anti-Clot Treatment Scale (ACTS) questionnaire to evaluate satisfaction related to oral anticoagulant treatment. The ACTS Burdens total score ranges from 12 to 60, and the ACTS Benefits total score ranges from 3 to 15. Higher ACTS Burdens and Benefits scores indicate greater satisfaction with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Peter Riber, DMSc, Principal Investigator — Odense University Hospital
Locations (6):
- Denmark (6):
  - Rigshospitalet, Copenhagen, Capital Region
  - Gentofte Hospital, Gentofte Municipality, Capital Region
  - Regionshospital Gødstrup, Herning, Central Jutland
  - Aalborg university hospital, Aalborg, North Denmark
  - Århus Universitetshospital, Aarhus, Region Midt
  - Odense University Hospital, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gosvig K, Goller J, Hansson NH, Brandes A, Modrau I, Rasmussen LF, Eskesen K, Jensen AKG, Belley-Cote E, Whitlock R, Riber LPS. Rationale and design of the anticoagulant therapy after left atrial appendage closure (ATLAAC) trial. Am Heart J. 2025 Sep;287:86-93. doi: 10.1016/j.ahj.2025.04.015. Epub 2025 Apr 15. PMID 40246048